CLINICAL TRIAL: NCT06162000
Title: Investigation of the Effect of Decision Support System Integrated Nursing Care Plan Management System on Student Nurses' Care Plan Preparation Skills
Brief Title: the Effect of Nursing Care Plan Management System on Student Nurses' Care Plan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Meltem ÖZDUYAN KILIÇ, Lecturer, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Meltem06Hacettepe
Record Dates: First submitted 2023-11-14; First posted 2023-12-08 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Nurse's Role
Keywords: Patient care plan; Decission Support System; Nursing Process; Nursing Education; Nursing Students

STUDY DESIGN:
Intervention Model Description: Posttest with control group
Who Masked: Outcomes Assessor
Masking Description: During the statistical analysis phase, codes as a and b will be given to the control and intervention groups and thus statistical bias will be controlled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group of nursing students (Experimental): The group that will use the developed software in case studies
  Interventions: Other: The group that will use the developed software in case studies
- Control Group of nursing students (No Intervention): Group that will prepare case studies on paper

INTERVENTIONS:
Other: The group that will use the developed software in case studies — In the study, a case study will be conducted with students in the control and intervention groups once a week for four weeks.
  Students in the control group will be given printed cases and asked to prepare care plans on ready-made paper templates.
  Case preparation activities of the students in the intervention group will be carried out in line with the software planned to be developed. Before the case preparation activities begin, an information/promotional meeting will be held regarding the use of the application planned to be developed. Students will log in to the application with their e-mail addresses and the password they will choose when they first log in. Students will be asked to review the software and questions regarding usage will be answered. Students will record patient data in the cases into KSDE-HBPYS and prepare care plans with the software. At the end of the case studies, a posttest case and Clinical Decision Making Scale will be applied to both groups.
  Arms: intervention group of nursing students

SUMMARY:
The goal of this post-test control group study is to evaluate the effect of the Clinical Decision Support Integrated Patient Care Plan Management System (KDSE-HBPYS) training tool on nursing students' ability to prepare a care plan and their perception of clinical decision-making.

Case studies will be conducted with control and intervention groups for 4 weeks. The paper based patient cases will give the students who is in the control group and they will prepare patients' care plans on the paper templates (template containing problem-related data, nursing diagnoses, purpose, outcome criteria, planning titles). Patient care preparation activities based on the cases will be carried out in line with the software with the intervention group. In the fifth week, students in both control and intervention groups will prepare a care pla for the final test case. At the conclusion of the final test case, students will be administered the Clinical Decision Making Scale.

The difference between the scores of students in the control and intervention groups from the post-test case and the scores they received from the clinical decision-making scale will be investigated.

DETAILED DESCRIPTION:
The significance of nursing care plans as tools for inter-professional communication within healthcare settings cannot be overstated. These care plans serve as comprehensive guides, not only to evaluate patient care outcomes but also to make transparent the nursing care process, thereby ensuring the delivery of high-quality and safe healthcare. Study findings underscore the impediments students encounter in fully integrating the nursing process into their patient care practices. Therefore, this study aims to evaluate the effect of the Clinical Decision Support Integrated Patient Care Plan Management System (KDSE-HBPYS) training tool on nursing students' ability to prepare a care plan and their perception of clinical decision-making.

Type of Research:

The research was planned as post-test control group study.

Research Hypotheses:

H0_1: Nursing process teaching through the Clinical Decision Support Integrated Patient Care Plan Management System (KDSE-HBPYS) increases students' ability to prepare a care plan.

H0_2: Nursing process teaching through the Clinical Decision Support Integrated Patient Care Plan Management System (KDSE-HBPYS) increases students' perception of clinical decision-making.

Population and Sample of the Research:

The population of the research will consist of second-year students studying at Ankara University Faculty of Nursing in the Fall Semester of the 2023-2024 Academic Year and agreeing to participate in the research. The power of the research will be calculated at the end of the study. Since students' academic achievement averages may affect the study results, stratified sampling method will be used to determine the control and intervention groups. Students who agree to participate in this study will be grouped according to their academic achievement averages, and then random assignment will be made to intervention and control groups. As the researcher must implement and evaluate the interventions, researcher blinding will not be possible. Since participants in the intervention group must use the application, participant blinding will not be possible. However, during the statistical analysis phase, codes as a and b will be given to the control and intervention groups, thus controlling statistical bias.

Criteria for Inclusion of the Control and Intervention Groups in the Research:

(i) Participated in theoretical and clinical teaching on the nursing process and preparation of a care plan within the Fundamentals of Nursing course.

Exclusion Criteria from the Study:

(i) Had taken the Internal Medicine Nursing Course in previous semesters, but not being successful in the course, (ii) Have been working as a nurse/nurse assistant/health officer etc. in any health institution.

Data Collection Forms

1. Personal Information Form
2. Nursing Care Plan Evaluation Case (posttest):
3. Clinical Decision Making Scale in Nursing

Application of Research:

In the study, the effectiveness of the Clinical Decision Support Integrated Patient Care Plan Management System (KDSE-HBPYS) will be evaluated.

KDSE-HBPYS is designed to allow planning the patient's care using the nursing process approach, recording the care practices performed, sharing them with the instructor and receiving feedback from the instructor. The data collection form used in the Fundamentals of Nursing Course in clinical teaching has been included in the design (data collection forms can be updated within the scope of the course to be used). In addition, standard assessment tools used in the patient's care; pain assessment form, nutrition assessment form, pressure sore assessment form, fall risk assessment form, etc. built into the design. While the research team was creating the content of the decision support system used the "Pearson Nursing Diagnoses Handbook" as a source which includes NANDA International (NANDA-I) Nursing Interventions Classification (NIC) and Nursing Outcomes Classification (NOC). The decision support system is a semi-active system which is automatically triggered and provides the user with information and recommendations based on standards/procedures regarding the current situation. In addition, international standards that decision support systems to be developed for the nursing process should meet were also used. In this direction, the first design of KSDE-HBPYS was carried out.

Implementation of the study and Collection of Data A meeting was made in order to inform students about the research and invite them to participate in the second week of the 2023-2024 Academic Year Fall Semester.

Students who agree to participate in the research were included in the study and their questions were answered. These students' contact information (name, surname, student number, telephone number) and their consent to participate in the research voluntarily were obtained, and an introductory information form were filled out. Then, they were assigned to control and intervention groups, and WhatsApp groups were created to maintain communication with students.

2023-2024 Academic Year Fall Semester, students will meet once a week for four weeks and a care plan will be prepared in line with the cases for which expert opinion has been received. In this context, researchers and students in both control and intervention groups will come together simultaneously in two separate classes within Ankara University Faculty of Nursing.

The cases will be given to the students in the control group in printed paper form and they will be asked to prepare their care plans on ready-made paper templates (on A4 paper; template containing problem-related data, nursing diagnoses, purpose, outcome criteria, planning titles). There will be no time limit for the student in the preparation of care plans. Any questions from students will be answered in order to provide students with a teaching experience similar to in clinical practice. Warning signs will be hung on the doors of the classrooms to prevent divisions during the application. Then, at the end of the case studies, the students will meet in a suitable classroom at Ankara University Faculty of Nursing on the determined day and time, and the students will prepare a care plan for the final test case. At the conclusion of the final test case, students will be administered the Clinical Decision Making Scale.

Case preparation activities of the students in the intervention group will be carried out in line with the software. Before the case preparation activities begin, an information/promotional meeting will be held on the use of the application. Students will log in to the application with their student numbers and the passwords they will choose when they first log in. Students will be asked to review the software and their questions regarding usage will be answered. The cases will be given to the students in paper forms, they will record the patients data in KSDE-HBPYS and they will prepare the care plans for the relevant case through the software. There will be no time limit for the student in the preparation of care plans. Warning signs will be hung on the doors of the classrooms to prevent divisions during the application. Then, at the end of the case studies, the students will meet in a suitable classroom at Ankara University Faculty of Nursing on the determined day and time, and the students will prepare a care plan for the final test case. At the conclusion of the final test case, students will be administered the Clinical Decision Making Scale.

ELIGIBILITY:
Inclusion Criteria:

* Participating in in-class theoretical and clinical teaching on the nursing process and preparation of a care plan within the Fundamentals of Nursing course.

Exclusion Criteria:

* Having taken the Internal Diseases Nursing Course in previous semesters, but not being successful in the course,
* She is a graduate of a health vocational high school and can work as a nurse/nurse assistant/health officer etc. in any health institution. It was determined as being working.

Ages: 19 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Nursing Care Plan Evaluation Case (post-test) Points | 1 week
  Nursing process teaching through the clinical support integrated patient care plan management system changes students' ability to prepare a care plan.
Clinical Decision Making Scale in Nursing (max:200 points, min: 40 points; higher scores mean a better outcome ) | 1 week
  Nursing process teaching through the decision support system integrated patient care plan management system changes students' perception of clinical decision-making.

CONTACTS AND LOCATIONS:
Overall Officials: FATOŞ KORKMAZ, PHD, Study Director — HACETTEPE UNIVERSİTY
Locations (1):
- Ankara University Faculty of Nursing, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parvan K, Hosseini FA, Jasemi M, Thomson B. Attitude of nursing students following the implementation of comprehensive computer-based nursing process in medical surgical internship: a quasi-experimental study. BMC Med Inform Decis Mak. 2021 Jan 6;21(1):10. doi: 10.1186/s12911-020-01378-6. PMID 33407383
- [Background] Ranjbar K, Sabetsarvestani R, Oghlaee H, Sarvestani PS, Dehghan A, Shirazi ZH. Using Electronic Software for Nursing Documentation in Nursing Students. Florence Nightingale J Nurs. 2021 Jun 1;29(2):128-136. doi: 10.5152/FNJN.2021.20077. eCollection 2021 Jun. PMID 34263231
- [Background] Warboys I, Mok WY, Frith KH. Electronic medical records in clinical teaching. Nurse Educ. 2014 Nov-Dec;39(6):298-301. doi: 10.1097/NNE.0000000000000072. PMID 25073041
- [Result] Muller-Staub M, de Graaf-Waar H, Paans W. An Internationally Consented Standard for Nursing Process-Clinical Decision Support Systems in Electronic Health Records. Comput Inform Nurs. 2016 Nov;34(11):493-502. doi: 10.1097/CIN.0000000000000277. PMID 27414705